CLINICAL TRIAL: NCT04261439
Title: A Phase I/Ib Study of Subcutaneous Recombinant Human NIZ985 ((hetIL-15) (IL-15/sIL-15Rα)) in Combination With Spartalizumab in Patients With Check Point Inhibitor (CPI) Relapsed Advanced Solid Tumors and Lymphoma
Brief Title: A Phase I/Ib Study of NIZ985 Alone and in Combination With Spartalizumab
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor's decision and not due to any safety concerns
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CNIZ985B12101; 2019-004069-42 (EudraCT Number)
Record Dates: First submitted 2020-02-06; First posted 2020-02-07 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: In Escalation: All Patients With Solid Tumors and Lymphoma; In Expansion: Melanoma, Non-small Cell Lung Cancer
Keywords: NIZ985; Spartalizumab; Tislelizumab; immunotherapy; checkpoint Inhibitor; checkpoint inhibitor resistance; melanoma; NSCLC
MeSH Terms: conditions — Lymphoma; Carcinoma, Non-Small-Cell Lung; Melanoma | interventions — spartalizumab; tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Single agent arm. NIZ985 is administered as a single agent (subjects may be treated with the NIZ985-Spartalizumab combination after their first disease re-evaluation)
  Interventions: Drug: NIZ985; Drug: Spartalizumab
- Arm 2 (Experimental): Combination arm. NIZ985 and Spartalizumab combination is administered starting at Cycle 1 Day 1 in dose escalation. NIZ985 and tislelizumab combination is administered starting at Cycle 1 Day 1 in dose expansion.
  Interventions: Drug: NIZ985; Drug: Spartalizumab; Drug: Tislelizumab

INTERVENTIONS:
Drug: NIZ985 — NIZ985 injection
Drug: Spartalizumab — Spartalizumab infusion
  Other Names: PDR001
Drug: Tislelizumab — Tislelizumab infusion
  Other Names: VDT482
  Arms: Arm 2

SUMMARY:
The purpose of this phase I/Ib study was to determine the safety profile of NIZ985 (new formulation), and if it could be safely combined with spartalizumab or tislelizumab and to determine the appropriate dose and schedule for further study. Moreover, the study characterized the pharmacokinetic profiles of NIZ985 as a single agent and in combination with spartalizumab or tislelizumab and identified preliminary anti-tumor activity.

DETAILED DESCRIPTION:
This was a phase I/Ib, open-label, global, multi-center study of subcutaneously administered NIZ985 alone and in combination with a PD-1 inhibitor in patients with advanced solid tumors and lymphoma who had progressed after obtaining a previous response to anti-PD-1/ CPI therapy at any time prior to enrollment. Previous response was defined as a radiographic complete response (CR) or a partial response (PR). Patients with stable disease (SD) lasting ≥ 6 months could also be included if the most recent regimen included CPI. The study consisted of two parts, dose escalation and dose expansion. Two separate arms were examined during the escalation portion: 1) evaluation of NIZ985 as a single agent. Spartalizumab could be added at the time of the first disease re-evaluation and 2) administration of NIZ985 and spartalizumab as a combination starting from C1D1. In dose expansion, NIZ985 was administered in combination with tislelizumab.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent must be obtained prior to participation in the study.
2. Male or female patients ≥ 18 years of age
3. Histologically confirmed and documented advanced solid tumors and lymphoma (includes locally advanced malignancies that are not curable by surgery or radiotherapy, and those with metastatic disease) with documented progression following standard therapy, and for whom, no standard therapy is available, tolerated or appropriate. Disease must be measurable as determined by RECIST 1.1 (refer to Appendix 1) or Cheson et al (2014) (refer to Appendix 6).

   * Escalation: Patients previously treated with CPI (anti PD-1/PD-L1 and/or anti CTLA-4) who have previously responded and progressed at any time prior to enrollment. Previous response is an initial radiographic CR/PR (a confirmatory scan is not required). If the most recent regimen included CPI, patients with SD lasting ≥ 6 months are also eligible.
   * Expansion in melanoma: Patients with cutaneous melanoma previously treated with CPI (anti PD 1/ PD-L1 and/or anti CTLA-4) who have previously responded and progressed at any time prior to enrollment. Previous response is radiographic CR/PR (a confirmatory scan is not required). If the most recent regimen included CPI, patients with SD lasting ≥ 6 months are also eligible.
   * Expansion in NSCLC: Patients with locally advanced or unresectable NSCLC who have been treated with up to 2 prior lines of therapies, at least one of which was a CPI-containing regimen (anti PD 1/ PD-L1 and/or anti CTLA-4). Patients must have previously responded to CPI and progressed at any time prior to enrollment. Previous response is radiographic CR/PR (a confirmatory scan is not required). If the most recent regimen included CPI, patients with SD lasting ≥ 6 months are also eligible. Patients with actionable mutations will be excluded.
4. Patients must be willing and able to comply with the protocol for the duration of the study
5. Patients must have a site of disease amenable to biopsy and be a candidate for tumor biopsy according to the treating institution's guidelines. Patient must be willing to undergo a new tumor biopsy at screening and during therapy on the study.
6. ECOG performance status ≤1 and in the opinion of the investigator, likely to complete at least 28 days of treatment.

Exclusion Criteria:

1. Patients that have received any prior IL-15 treatment.
2. History of severe hypersensitivity reactions to any ingredient of study drug(s) and other mAbs and/or their excipients. In addition, patients with a history of immune mediated toxicities from CPI that led to permanent discontinuation of CPI treatment will be excluded.
3. Patients with primary CNS tumors are excluded. Presence of symptomatic CNS metastases, or CNS metastases that require local CNS-directed therapy (such as radiotherapy or surgery), or increasing doses of corticosteroids 2 weeks prior to study entry. Patients with treated symptomatic brain metastases should be neurologically stable (for 4 weeks post-treatment and prior to study entry) and at a dose of ≤ 10 mg per day prednisone or equivalent for at least 2 weeks before administration of any study treatment.
4. Systemic chronic steroid therapy (> 10mg/day prednisone or equivalent) or any immunosuppressive therapy, other than replacement-dose steroids in the setting of adrenal insufficiency, within 7 days of the first dose of study treatment. Topical, inhaled, nasal and ophthalmic steroids are allowed.
5. Malignant disease, other than that being treated in this study, that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer or other tumors that will not affect life expectancy.
6. Patients having out of range lab values during screening and before the first dose of study treatment. Out of range lab values are defined as:

   * Absolute neutrophil count (ANC) <1.0 x 109/L
   * Platelets <75 x 109/L
   * Hemoglobin (Hgb) < 9 g/dL
   * Serum creatinine > 1.5 x ULN or creatinine clearance < 60mL/min using Cockcroft-Gault formula (See Appendix 3)
   * Total bilirubin > 1.5 x ULN, (except for patients with Gilbert's syndrome > 3.0 x ULN or direct bilirubin > 1.5 x ULN)
   * Aspartate transaminase (AST) > 3 x ULN
   * Alanine transaminase (ALT) > 3x ULN
   * Serum electrolytes ≥ grade 2 despite adequate supplementation.
7. Impaired cardiovascular function or clinically significant cardiovascular disease, including any of the following:

   * Clinically significant and/or uncontrolled heart disease such as congestive heart failure requiring treatment (NYHA Grade ≥ 2), uncontrolled hypertension or clinically significant arrhythmia
   * QTcF >470 msec on screening ECG or congenital long QT syndrome
   * Acute myocardial infarction or unstable angina < 3 months prior to study entry
8. Infection(s):

   * HIV infection
   * Active HBV or HCV infection (per institutional guidelines). Patients with chronic HBV or HCV disease that is controlled under antiviral therapy are allowed in expansion but not in escalation.
   * Documented infection. Patients requiring systemic antibiotics for infection must have completed treatment before screening is initiated.
9. Active, known or suspected autoimmune disease. Patients with vitiligo, type I diabetes, residual hypothyroidism only requiring hormone replacement, psoriasis not requiring systemic treatment or conditions not expected to recur may be considered. Patients previously exposed to CPI treatment who were adequately treated for skin rash or with replacement therapy for endocrinopathies should not be excluded.
10. History of or current interstitial lung disease or pneumonitis grade ≥ 2.
11. Radiotherapy within 2 weeks of the first dose of study drug, except for palliative radiotherapy to a limited field. To allow evaluation for response to study treatment, patients enrolled in the expansion must have remaining measurable disease that has not been irradiated.
12. Treatment with cytotoxic or targeted antineoplastics within 3 weeks of initiation of study treatment. For cytotoxic agents that have major delayed toxicities, a washout period of one cycle is indicated (examples are nitrosoureas and mitomycin C which typically require a 6 week washout). Prior antibodies or immunotherapies require a 4 week washout. Ongoing bisphosphonate therapy and growth hormone-releasing hormone (GHRH) agonist therapy is allowed. Supportive therapy with denosumab is allowed. For patients with lymphoma, the following washout criteria may be used:

    • Systemic antineoplastic therapy (including cytotoxic chemotherapy, alfa-interferon, kinase inhibitors or other targeted small molecules, and toxin immunoconjugates) or any experimental therapy within 14 days or 5 half-lives, whichever is shorter, before the first dose of study treatment
13. Presence of Grade ≥ 2 toxicity according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE v5.0), from prior cancer therapy with the exception of neuropathy (inclusion of patients with neuropathy of Grade 2 or less is permitted), ototoxicity, and alopecia.
14. Two weeks since major surgery treatment (mediastinoscopy, insertion of a central venous access device and insertion of a feeding tube are not considered major surgery)
15. Use of any live vaccines against infectious diseases within 4 weeks of initiation of study treatment.
16. Use of hematopoietic growth factors or transfusion support ≤ 2 weeks prior to start of study treatment. If growth factors were initiated more than 2 weeks prior to the first dose of study treatment and the patient is on a stable dose, they can be maintained.
17. Any medical condition that would, in the investigator's judgement, prevent the patient's participation in the clinical study due to safety concerns, compliance with clinical study procedures, or interpretation of study results.
18. Pregnant or nursing (lactating) women.
19. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception while taking study medication and for 30 days after the last dose of NIZ985 if receiving NIZ985 alone, 120 days after last dose of tislelizumab, or for 150 days after the last dose of spartalizumab. Highly effective methods of contraception methods include:

    * Total abstinence (when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
    * Female bilateral tubal ligation, female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or total hysterectomy at least six weeks before taking investigational drug(s). In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
    * Male sterilization (at least 6 months prior to screening). For female patients on the study, the vasectomized male partner should be the sole partner for that patient
    * Use of oral (estrogen and progesterone), injected, or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS), or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example, hormone vaginal ring or transdermal hormone contraception.
    * In case of use of oral contraception women should have been stable on the same pill for a minimum of 3 months before taking study treatment.

    NOTE: Women are considered post-menopausal and not of child-bearing potential if they have had over 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate [generally age from 40 to 59 years], history of vasomotor symptoms [e.g. hot flush]) in the absence of other medical justification or have had surgical bilateral oophorectomy (with or without hysterectomy), total hysterectomy or bilateral tubal ligation at least six weeks prior to enrollment on study. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child-bearing potential.
20. A condom is required for all sexually active male participants to prevent them from fathering a child AND to prevent delivery of study treatment via seminal fluid to their partner. Sexually active males receiving NIZ985 as a single agent or in combination with spartalizumab or tislelizumab must use a condom during intercourse for 30 days after their last dose of NIZ985. In addition, male participants must not donate sperm for 30 days after the last dose of NIZ985. Patients should not father a child during this post treatment period. A condom is required to be used also by vasectomized men as well as during intercourse with a male partner in order to prevent delivery of the drug via semen.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-02-27 (Actual); Primary Completion 2023-12-27 (Actual); Study Completion 2023-12-27 (Actual)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxcities (DLTs) in escalation and expansion | 1 cycle (28 days)
  Incidence of DLTs in Cycle 1 (28 days) in escalation and expansion
Number of patients with and severity of adverse events (AEs) and serious adverse events (SAEs) | 24 months
  AEs and SAEs including changes in laboratory parameters, vital signs and electrocardiograms (ECGs) qualifying and reported as AEs for all patients from escalation and expansion
Dose interruptions and reductions | 24 months
  Number of dose interruptions and dose reductions of NIZ985, spartalizumab and tislelizumab.
Dose intensity | 24 months
  Dose intensity as a ratio of cumulative dose received during duration of exposure over duration of exposure for NIZ985, spartalizumab and tislelizumab.

SECONDARY OUTCOMES:
Overall response Rate (ORR) | 24 months
  as per RECIST 1.1 or Cheson (2014)
Best Overall Response (BOR) | 24 months
  as per RECIST1.1 or Cheson (2014)
Disease control Rate (DCR) | 24 months
  as per RECIST 1.1 or Cheson (2014)
Progression Free Survival (PFS) (expansion groups only) | 24 months
  as per RECIST 1.1 or Cheson (2014)
Duration of Response (DOR) (expansion groups only) | 24 months
  as per RECIST 1.1 or Cheson (2014)
Pharmacokinetics (PK) of NIZ985 (as a single agent and in combination), spartalizumab (in combination), and tislelizumab (in combination) | 24 months
  Measurement of serum concentrations of NIZ985, spartalizumab, and tislelizumab
Prevalence and incidence of immunogenicity of NIZ985 (single agent and in combination), spartalizumab (in combination), or tislelizumab (in combination) | 24 months
  Measurement of serum antidrug antibodies (ADA) to NIZ985, spartalizumab, and tislelizumab at baseline and on treatment

CONTACTS AND LOCATIONS:
Locations (9):
- United States (2):
  - City of Hope National Medical, Duarte, California
  - Moores UCSD Cancer Center, La Jolla, California
- Novartis Investigative Site, Leuven, Belgium
- Novartis Investigative Site, Essen, Germany
- Novartis Investigative Site, Napoli, Italy
- Novartis Investigative Site, Chuo Ku, Tokyo, Japan
- Spain (2):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study Results — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18219
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2412